CLINICAL TRIAL: NCT01987232
Title: Phase 1b/2, Multicenter, Open-label Study of Carfilzomib, Carboplatin, and Etoposide in Subjects With Previously Untreated Extensive-stage Small-cell Lung Cancer
Brief Title: Phase 1b/2 Study of Carfilzomib, Carboplatin, and Etoposide in Patients With Previously Untreated Extensive Stage Small-cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CFZ004; 2013-002597-44 (EudraCT Number); 20130399 (Other: Amgen Inc.)
Record Dates: First submitted 2013-11-06; First posted 2013-11-19 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Extensive-Stage Small-Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — carfilzomib; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib Combination (Experimental): Participants received carfilzomib on days 2, 3, 9, and 10 of each 21-day cycle as per the dose escalation schema, carboplatin at a target area under the curve (AUC) of 5 on day 1 of each cycle, and etoposide 100 mg/m² on days 1, 2, 3 of each 21-day cycle for up to 6 cycles. Participants with stable disease or better continued to receive carfilzomib alone until progressive disease (PD), unacceptable toxicity, withdrawal of consent, study closure, or death, whichever occurred earliest.
  Interventions: Drug: Carfilzomib; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Carfilzomib — Administered by intravenous infusion.
  Other Names: PR-171; PR171; Kyprolis®
Drug: Carboplatin — Administered by intravenous infusion.
Drug: Etoposide — Administered by intravenous infusion.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and assess the safety, tolerability and activity of carfilzomib given in combination with carboplatin and etoposide as initial therapy for patients with extensive-stage small-cell lung cancer (ES SCLC).

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of extensive-stage small-cell lung cancer (ES-SCLC) with measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1; ES-SCLC is defined as: small-cell lung cancer (SCLC) that has spread beyond one hemithorax and regional lymph nodes on the same side (e.g., supraclavicular) to the contralateral hemithorax, lymph nodes, or more distant locations in the body
2. Subjects with asymptomatic brain metastases or other central nervous system (CNS) disease at screening/diagnosis are eligible
3. Males and females ≥ 18 years of age
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Key Exclusion Criteria:

1. Previous systemic therapy to treat small-cell lung cancer (SCLC). Subjects with recurrent or progressive limited-stage SCLC after previous systemic treatment are not eligible for study participation.
2. Whole brain or focal radiation therapy within 14 days prior to Cycle 1 Day 1 (C1D1) for Phase 1b or prior to randomization for Phase 2
3. Congestive heart failure (New York Heart Association [NYHA] class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months prior to prior to C1D1 for Phase 1b or prior to randomization for Phase 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-11-05; Primary Completion 2016-08 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- United States (11):
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - UF Health Davis Cancer Pavilion and Shands Med Plaza, Gainesville, Florida
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana
  - Baptist Health Lexington Clinical Research Center, Lexington, Kentucky
  - Frederick Memorial Hospital, Frederick, Maryland
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Juravinski Cancer Centre, Hamilton, Ontario, Canada
- Russia (5):
  - Regional Budgetary Healthcare Institution "Kursk Regional Clinical Oncology Dispensary", Kislino, Kursk Oblast
  - State budgetary healthcare institution of Arkhangelsk Region "Arkhangelsk Clinical Oncological Dispensary", Arkhangelsk
  - Federal State Budgetary Scientific Institution "N.N. Blokhin Russian Cancer Research Center", Moscow
  - State Budgetary Educational Inslitution of Higher Professional Education "First St. Petersburg I.P.Pavlov State Medical University", Saint Petersburg
  - State Budgetary Healthcare Institution of Yaroslavl Region "Regional Clinical Oncological Hospital", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 17 centers in the United States, Russia, and Canada.
Pre-assignment Details: In the phase 1b portion of the study participants were assigned sequentially to escalating doses of carfilzomib given in combination with standard dose carboplatin and etoposide to establish the maximum tolerated dose (MTD). The phase 2 portion of the study was not enrolled.
Groups:
- Carfilzomib 20/20 mg/m²: Participants received carfilzomib 20 mg/m² on days 2, 3, 9, and 10 of each 21-day cycle, carboplatin at a target area under the curve (AUC) of 5 on day 1 of each cycle, and etoposide 100 mg/m² on days 1, 2, and 3 of each 21-day cycle for up to 6 cycles. Participants with stable disease or better continued to receive carfilzomib alone until progressive disease (PD), unacceptable toxicity, withdrawal of consent, study closure, or death, whichever occurred earliest.
- Carfilzomib 20/27 mg/m²: Participants received carfilzomib 20 mg/m² on cycle 1 days 2 and 3, then 27 mg/m² on days 9 and 10 and thereafter for each subsequent 21-day cycle, carboplatin at a target AUC of 5 on day 1 of each cycle, and etoposide 100 mg/m² on days 1, 2, and 3 of each cycle for up to 6 cycles. Participants with stable disease or better continued to receive carfilzomib alone until PD, unacceptable toxicity, withdrawal of consent, study closure, or death, whichever occurred earliest.
- Carfilzomib 20/36 mg/m²: Participants received carfilzomib 20 mg/m² on cycle 1 days 2 and 3, then 36 mg/m² on days 9 and 10 and thereafter for each subsequent 21-day cycle, carboplatin at a target AUC of 5 on day 1 of each cycle, and etoposide 100 mg/m² on days 1, 2, and 3 of each cycle for up to 6 cycles. Participants with stable disease or better continued to receive carfilzomib alone until PD, unacceptable toxicity, withdrawal of consent, study closure, or death, whichever occurred earliest.
- Carfilzomib 20/45 mg/m²: Participants received carfilzomib 20 mg/m² on cycle 1 days 2 and 3, then 45 mg/m² on days 9 and 10 and thereafter for each subsequent 21-day cycle, carboplatin at a target AUC of 5 on day 1 of each cycle, and etoposide 100 mg/m² on days 1, 2, and 3 of each cycle for up to 6 cycles. Participants with stable disease or better continued to receive carfilzomib alone until PD, unacceptable toxicity, withdrawal of consent, study closure, or death, whichever occurred earliest.
- Carfilzomib 20/56 mg/m²: Participants received carfilzomib 20 mg/m² on cycle 1 days 2 and 3, then 56 mg/m² on days 9 and 10 and thereafter for each subsequent 21-day cycle, carboplatin at a target AUC of 5 on day 1 of each cycle, and etoposide 100 mg/m² on days 1, 2, and 3 of each cycle for up to 6 cycles. Participants with stable disease or better continued to receive carfilzomib alone until PD, unacceptable toxicity, withdrawal of consent, study closure, or death, whichever occurred earliest.
Period: Overall Study
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m²
Started | 5 | 3 | 3 | 15 | 6
Completed | 5 | 3 | 3 | 14 | 6
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Ongoing in Study | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Carfilzomib 20/20 mg/m²: Participants received carfilzomib 20 mg/m² on days 2, 3, 9, and 10 of each 21-day cycle, carboplatin at a target AUC of 5 on day 1 of each cycle, and etoposide 100 mg/m² on days 1, 2, and 3 of each 21-day cycle for up to 6 cycles. Participants with stable disease or better continued to receive carfilzomib alone until PD, unacceptable toxicity, withdrawal of consent, study closure, or death, whichever occurred earliest.
- Total: Total of all reporting groups
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m² | Total
Number analyzed (Participants) | 5 | 3 | 3 | 15 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (13.8) | 62.3 (8.5) | 59.0 (7.5) | 56.9 (9.4) | 58.8 (7.9) | 59.9 (10.1)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 2 | 2 | 2 | 14 | 5 | 25
  ≥ 65 years | 3 | 1 | 1 | 1 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 5 | 1 | 12
  Male | 2 | 1 | 2 | 10 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 3 | 3 | 14 | 5 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 3 | 3 | 14 | 6 | 31
  Other | 0 | 0 | 0 | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active; 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, no self-care, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 4 | 0 | 1 | 3 | 2 | 10
    1 (Restrictive but ambulatory) | 1 | 3 | 2 | 12 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities
Description: The maximum tolerated dose (MTD) was defined as the highest dose level at which < 33% of participants experienced a dose-limiting toxicity (DLT) during the first 21-day cycle. Dose-limiting toxicities were evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03. A DLT was defined as:
  * A grade 3 or greater non-hematologic toxicity that was assessed as related to carfilzomib by the investigator except in the case of neuropathy. A grade 2 or higher neuropathy with pain was considered a DLT.
  * Grade 4 neutropenia: absolute neutrophil count (ANC) < 500 mm³, lasting ≥ 7 days despite granulocyte colony stimulating factor support, or any febrile (temperature > 38.3°C) neutropenia (ANC < 1000 mm³).
  * Thrombocytopenia of any grade associated with clinically significant bleeding or platelet/blood transfusion
  * Grade 4 fatigue lasting ≥ 7 days
  * Grade 3 nausea, vomiting or diarrhea lasting ≥ 7 days.
Time Frame: First 21-day Cycle
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m²
Number analyzed (Participants) | 5 | 3 | 3 | 15 | 6
Participants | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The severity of each adverse event was assessed using the NCI-CTCAE Version 4.03 according to the following:
  Grade 1 - Mild: Asymptomatic or mild symptoms; intervention not indicated
  Grade 2 - Moderate: Minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)
  Grade 3 - Severe: Medically significant but not life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL
  Grade 4 - Life-threatening
  Grade 5 - Fatal.
  A serious AE is an AE that met one or more of the following criteria:
  * Death
  * Life-threatening
  * Required inpatient hospitalization or prolongation of an existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * A congenital anomaly/birth defect
  * Important medical events that required medical or surgical intervention to prevent one of the outcomes above.
Time Frame: From first day of any study treatment (i.e., carfilzomib, carboplatin, or etoposide) up to 30 days after the last day of study treatment. The median overall duration of treatment was 16 weeks.
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m²
Number analyzed (Participants) | 5 | 3 | 3 | 15 | 6
Participants
  Any adverse event | 5 | 3 | 3 | 15 | 5
  Adverse events ≥ grade 3 | 3 | 3 | 2 | 13 | 4
  Serious adverse events | 1 | 1 | 1 | 7 | 2
  AEs leading to disocontinuation of study drug | 1 | 0 | 0 | 3 | 1
  Fatal adverse events | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: Overall Survival (OS) - Phase 2
Description: Overall Survival (OS) is defined as the time from randomization to the date of death. Overall survival was a specified secondary endpoint for the phase 2 portion of the study; since phase 2was not conducted, OS was not analyzed.
Time Frame: 30 months
Population: Participants enrolled in phase 2
Groups:
- All Participants: Participants received carfilzomib on days 2, 3, 9, and 10 of each 21-day cycle, carboplatin at a target AUC of 5 on day 1 of each cycle, and etoposide 100 mg/m² on days 1, 2, and 3 of each 21-day cycle for up to 6 cycles. Participants with stable disease or better continued to receive carfilzomib alone until PD, unacceptable toxicity, withdrawal of consent, study closure, or death, whichever occurred earliest.
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m² | All Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Maximum Plasma Concentration - Phase 2
Description: Pharmacokinetic (PK) analyses were specified as secondary endpoints for the phase 2 portion of the study; since phase 2 was not conducted, PK analyses were not performed.
Time Frame: Cycle 1 Day 2
Population: Phase 2 participants
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m² | All Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Time of Maximum Plasma Concentration - Phase 2
Description: as for outcome 4
Time Frame: Cycle 1 Day 2
Population: Phase 2 participants
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m² | All Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Area Under Plasma Concentration-Time Curve - Phase 2
Description: as for outcome 4
Time Frame: Cycle 1 Day 2
Population: Phase 2 participants
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m² | All Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Other Pre Specified Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was specified as a primary endpoint for the phase 2 portion of the study. Since phase 2 did not proceed PFS was analyzed in phase 1b participants on an exploratory basis. PFS was defined as the time from the start of treatment to documented disease progression or death due to any cause, whichever occurred first. Disease progression was determined by the investigator according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, defined as at least a 20% increase in the size of target lesions (absolute increase ≥ 5 mm), unequivocal progression of existing non-target lesions, or any new lesions.
  Median PFS was calculated using Kaplan-Meier methods. Participants with no baseline disease assessments, who started a new anticancer therapy before documentation of PD or death, with death or PD immediately after more than 1 consecutively missed disease assessment visit or alive without documentation of PD before the data cutoff date were censored.
Time Frame: From first dose of study drug until the end of treatment; median duration of treatment was 16 weeks.
Population: All participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m² | All Participants
Number analyzed (Participants) | 5 | 3 | 3 | 15 | 6 | 32
months | 4.0 [2.8 to 6.7] | 6.4 [6.2 to 6.8] | 7.0 [4.0 to 7.0] | 2.9 [2.5 to 5.4] | 3.8 [1.1 to 6.3] | 4.4 [2.8 to 5.6]

8. Other Pre Specified Outcome: Overall Response Rate
Description: The overall response rate (ORR) was defined as the percentage of participants for whom the best overall confirmed response was either complete response (CR) or partial response (PR) assessed by the investigator according to RECIST v1.1 criteria.
  CR: Disappearance of all target and non-target lesions, no new lesions and normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters, or, the disappearance of all target lesions and persistence of one or more non-target lesion(s) and/or maintenance of tumor marker levels above normal limits.
Time Frame: From first dose of study drug until the end of treatment; median duration of treatment was 16 weeks.
Population: All participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: Participants received carfilzomib on days 2, 3, 9, and 10 of each 21-day cycle, carboplatin at a target area AUC of 5 on day 1 of each cycle, and etoposide 100 mg/m² on days 1, 2, and 3 of each 21-day cycle for up to 6 cycles. Participants with stable disease or better continued to receive carfilzomib alone until PD, unacceptable toxicity, withdrawal of consent, study closure, or death, whichever occurred earliest.
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m² | All Participants
Number analyzed (Participants) | 5 | 3 | 3 | 15 | 6 | 32
percentage of participants | 60.0 [14.7 to 94.7] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2] | 33.3 [11.8 to 61.6] | 33.3 [4.3 to 77.7] | 46.9 [29.1 to 65.3]

9. Other Pre Specified Outcome: Duration of Response
Description: Duration of response (DOR) was calculated for participants who achieved a confirmed CR or PR. defined as the time from first evidence of confirmed PR/CR to disease progression or death due to any cause. Median DOR was calculated using Kaplan-Meier methods. Participants with no baseline disease assessments, who started a new anticancer therapy before documentation of PD or death, with death or PD immediately after more than 1 consecutively missed disease assessment visit or alive without documentation of PD before the data cutoff date were censored.
  DOR was originally specified as a secondary endpoint for the phase 2 portion of the study. Since phase 2 did not proceed, DOR was analyzed in phase 1b participants on an exploratory basis.
Time Frame: From first dose of study drug until the end of treatment; median duration of treatment was 16 weeks.
Population: Participants with a confirmed response of PR or CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m² | All Participants
Number analyzed (Participants) | 3 | 3 | 2 | 5 | 2 | 15
months | 4.9 [2.8 to 5.4] | 5.0 [4.7 to 5.6] | NA [2.8 to NA] — Could not be estimated due to the low number of events | 4.3 [1.6 to NA] — Could not be estimated due to the low number of events | 4.5 [4.2 to 4.8] | 4.8 [2.8 to 5.4]

ADVERSE EVENTS:
Time Frame: From first day of any study treatment (i.e., carfilzomib, carboplatin, or etoposide), and within 30 days of the last day of study treatment. The median overall duration of treatment was 16 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Carfilzomib 20/27 mg/m²: Participants received carfilzomib 20 mg/m² on cycle 1 days 2 and 3, then 27 mg/m² on days 9 and 10 and thereafter for each subsequent 21-day cycle, carboplatin at a target AUC of 5 on day 1 of each cycle, and etoposide 100 mg/m² on days 1, 2, and 3 of each cycle for up to 6 cycles. Participants with stable disease or better continued to receive carfilzomib alone until progressive disease (PD), unacceptable toxicity, withdrawal of consent, study closure, or death, whichever occurred earliest.
Arm/Group | Carfilzomib 20/20 mg/m² | Carfilzomib 20/27 mg/m² | Carfilzomib 20/36 mg/m² | Carfilzomib 20/45 mg/m² | Carfilzomib 20/56 mg/m²
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/3 | 1/3 | 7/15 | 2/6
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 3/3 | 15/15 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib 20/20 mg/m² (N=5) | Carfilzomib 20/27 mg/m² (N=3) | Carfilzomib 20/36 mg/m² (N=3) | Carfilzomib 20/45 mg/m² (N=15) | Carfilzomib 20/56 mg/m² (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Injection site abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib 20/20 mg/m² (N=5) | Carfilzomib 20/27 mg/m² (N=3) | Carfilzomib 20/36 mg/m² (N=3) | Carfilzomib 20/45 mg/m² (N=15) | Carfilzomib 20/56 mg/m² (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 8 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 10 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 7 | 4
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 5 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 3 | 5 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 2 | 1
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 4 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 2 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Injection site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Incision site swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 1 | 2
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 2 | 0 | 1 | 1 | 2
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 2 | 0 | 2 | 2
Weight decreased (Investigations) | 0 | 0 | 1 | 2 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Decreased vibratory sense (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 3 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 2 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Hyporeflexia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 5 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.